CLINICAL TRIAL: NCT03454009
Title: Kent State University / Price Chopper Wellness Promotion Study
Brief Title: Kent State University / Price Chopper Employee Wellness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: The Golub Corporation, Price Chopper / Market 32 (Unknown); Cascades Tissue Group (Unknown)
Responsible Party: Principal Investigator, Maggie Stedman-Smith, Assistant Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-052
Record Dates: First submitted 2018-02-22; First posted 2018-03-05 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Acute Respiratory Infection; Influenza-like Illness; Gastrointestinal Infection
Keywords: multi-modal intervention;; office-based employees; hand hygiene; hand sanitizer; hand sanitizer surface wipes; self-reported infections; absenteeism; presenteeism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal hygiene intervention (Experimental): Employees will receive hygiene supplies including hand sanitizer, hand sanitizer surface disinfectant wipes and tissues, along with the following educational materials: a 2-minute electronic educational video; weekly 30-second electronic videos; and an educational flyer. Training materials discuss the importance of performing hygiene behaviors to prevent the spread of pathogens, such as, cleaning hands, using tissues to cover one's mouth and nose when coughing or sneezing, and keeping office surfaces clean.
  In addition, hygiene materials will be placed in common areas frequented by employees in the intervention group that include, educational hygiene posters, free standing hand sanitizer delivery stands, and bottles of hand sanitizer .
  Interventions: Behavioral: Multimodal hygiene intervention
- Control (No Intervention): Employees will complete all surveys but will not have access to additional hygiene products. Will follow usual hygiene behaviors.

INTERVENTIONS:
Behavioral: Multimodal hygiene intervention — hygiene supplies including hand sanitizer, hand sanitizer surface disinfectant wipes and tissues, along with the following educational materials: a 2-minute electronic educational video; weekly 30-second electronic videos; and an educational flyer.
  Arms: Multimodal hygiene intervention

SUMMARY:
This is a comprehensive randomized cluster hand-hygiene improvement intervention to reduce: self-reported acute respiratory tract infections (ARI) / influenza-like-illness (ILI) and gastrointestinal (GI) illness, absenteeism, presenteeism; and related behavioral and attitudinal change over a 90 day trial. The Intervention group will receive hand hygiene supplies, and a variety of educational materials, including environmental posters in common areas. The control group will perform their usual hygiene activities and will not receive an intervention.

Identical weekly surveys will be administered to the intervention and control groups to measure self-reported illness, absenteeism, presenteeism, along with behavior and attitudes measured at specified intervals during the study. The intervention and control groups were randomized by work floors before the onset of the enrollment period. It is hypothesized that employees in the intervention group will experience reduced self-reported illness, absenteeism and presenteeism along with improved protective hygiene behaviors and related attitudes, relative to those in the control group over the 90-day trial.

DETAILED DESCRIPTION:
The annual costs of seasonal influenza in the United States have been estimated at $87.1 billion, while costs from the common cold have been estimated at $40 billion. Office employees are at increased risk for contracting communicable disease at work, since they spend nearly half of their waking hours in this setting, work in close proximity with each other, and share equipment. Furthermore, employers in the U.S. have a compelling interest to reduce the spread of infectious disease, because they pay for the direct and indirect costs of absenteeism in employee wages, replacement of staff, reduced quality of services, rising health care premiums, and if self-insured, direct health care expenditures.

Hand hygiene is the single most important action to reduce the transmission of pathogens that result in healthcare acquired infections. Moreover, hand hygiene and respiratory etiquette have been recommended as primary non-pharmaceutical strategies in the early stages of an epidemic before a suitable vaccine is available. While influenza vaccine uptake is the most important recommendation to prevent influenza, the vaccine only protects against 3 or 4 of the most prevalent circulating strains in a given flu season and does not provide protection against non-influenza viral and bacterial pathogens. Meta-analysis has shown that numerous community intervention studies in schools, daycare, and private homes have reduced illness from infectious disease by 21-31%.

Despite the enormous burdens from communicable disease and the importance of the workplace as a setting for the potential spread of infections, to date, only four randomized control trials have been performed world-wide among office-based employees to assess the efficacy of hand hygiene interventions to reduce the spread of communicable disease, including acute respiratory infections (ARI), influenza-like illness (ILI) and gastrointestinal infections. Collectively, these interventions have shown promising results. Hubner and colleagues (2010) found a 65% reduction in the odds of contracting the common cold among workers with improved hand hygiene in a public administrative setting in Germany while Savolainen-Kopra and colleagues (2012) found a reduction in infectious illness among office employees in Finland who participated in a study arm that utilized soap and water and educational training. In the U.S., Stedman-Smith and colleagues (2015) found a 31% significant reduction in self-reported ARI / ILI and gastrointestinal illness combined in a multi-modal hand hygiene pilot randomized cluster trial among office employees at a Midwestern government center. While, Arbogast and colleagues (2016) found a significant reduction in health care claims for communicable infections spread by hand-to-mouth modes of transmissions over a 13-month, multi-component hand hygiene trial which utilized education, hand sanitizer and disinfectant wipes.

This is a comprehensive non-pharmaceutical randomized cluster hygiene improvement intervention to reduce self-reported acute respiratory tract infections (ARIs) / influenza-like-illness (ILI) and gastrointestinal (GI) illness, absenteeism, and presenteeism over a 90-day trial. The Intervention group will receive hygiene supplies (hand sanitizer, surface disinfectant wipes, tissues) and educational materials in varied mediums, including brief educational videos, and motivational posters hung in common work areas, in addition to hand sanitizer, along with hand sanitizer and surface disinfectant wipes installed in shared work areas. The control group will perform their usual hygiene activities and will not receive an intervention. Predominate pathways for the spread of ARI/ILI and non-foodborne GI infections include: (1) droplets that land on the nose, mouth, or are inhaled from infected persons' who cough, sneeze or talk; or (2) pathogens on hands contaminated from fomites or from touching infected persons, which come in contact with portals of entry including the mouth and nose. This multi-modal intervention is developed to promote improvements in the performance of protective behaviors that will reduce the spread of pathogens for ARI/ILI and GI infections by minimizing exposure from these two common pathways.

Identical weekly surveys will be administered to the intervention and control groups to measure self-reported illness, absenteeism and presenteeism; related behavior and attitudinal beliefs will be included in the surveys at specified longer intervals during the study. A sub-analysis will be performed to determine if those at high-risk for complications resulting in severe morbidity and mortality from infections show a reduction in self-reported infections, absenteeism and presenteeism. The intervention and control groups were randomized by work floors before the onset of the enrollment period.

It is hypothesized that employees in the intervention group will experience reduced self-reported illness, absenteeism and presenteeism along with improved protective hygiene behaviors, and attitudinal beliefs relative to those in the control group over the 90-day trial. Statistical analysis will be performed to determine if a relative reduction in self-reported communicable infections, absenteeism, and presenteeism, along with the improvement of related behaviors and attitudinal beliefs occurred among members in the intervention group relative to the control group over the 90-day trial. Statistical analysis will include the use of multiple imputation to impute missing variables, and the calculation of incidence rate ratios with 95% confidence intervals. Incident rate ratios will be calculated using generalized linear mixed models with a Poisson distribution and a log link function that will be adjusted for potential confounders and intercluster correlation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older
* No known allergies to alcohol or surface disinfecting wipes;
* Works at least 30% of office hours at the study host site;
* Consent to receiving emails from Kent State University.

Exclusion Criteria:

* Under 18 years of age;
* Known allergies to alcohol or surface disinfecting wipes;
* Works less than 30% of office hours at the study host site;
* Does not consent to receiving emails from Kent State University.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Reduction in ARI/ILI/GI infections as Self-Reported in Questionnaire | Approximately 90 days
  The content in this measurement item has demonstrated acceptable validity and reliability in a previous study from a scale that does not have a formal title, utilized by Stedman-Smith, DuBois and Grey (2012). The scale measures whether or not participants have had self-reported (1) acute respiratory tract / influenza-like infections (ARI/ILI) or (2) gastrointestinal (GI) infections with definitions used from the Centers for Disease Control and Prevention (CDC). Measurements will occur baseline, and once per week for 12 successive weeks until the end of the trial. The number of all self-reported infections during the 3-month trial will be counted, combined and summed in the intervention and the control groups; each sum will be used to compute incidence rates and an incidence rate ratio with a 95% confidence interval (CI).
Reduction in Absenteeism as Self-Reported in Questionnaire | Approximately 90 days
  Survey measurements will occur at baseline, and once per week for 12 successive weeks until the end of the trial. The content in this measurement item has demonstrated acceptable validity and reliability in a previous study from a scale that does not have a formal title, utilized by Stedman-Smith, DuBois and Grey (2012). The item contains a 6-point scale from zero days lost (0) to more than 5 days lost (6). The question was slightly adapted to add the response option of missing ½ day of work. The total number of lost work-days will be counted and summed from the 12 weekly surveys in the intervention and control group. Incidence rates and an incidence rate ratio with a 95% confidence interval will be calculated. Person days observed for this measurement will exclude holidays and weekends to match the intent of the survey regarding missed scheduled work-days.
Reduction in Presenteeism as Self-Reported in Questionnaire | Approximately 90 days
  Survey measurements will occur at baseline and once per week for 12 successive weeks until the end of the trial. This measurement is based upon 3 items on the Stanford Presenteeism Scale (SPS). Each of the 3 items are measured on a scale of 1-5 points from strongly agree (1 point) to strongly disagree (5 points). The original SPS construct measured these same items from a scale of strongly disagree to strongly agree; we have modified this in order to be consistent with the order of the rest of the questions in our survey, which range from positive to negative responses. The higher the number of points, the greater the degree of presenteeism (symptoms of illness while working). The mean score for presenteeism will be calculated in the intervention and control groups; the mean differences in the two groups will be compared, along with a 95% CI.

SECONDARY OUTCOMES:
Reduction in ARI/ILI/GI Infections among those at Highest Risk for Complications as Self-Reported in Questionnaire | Approximately 90 days
  Analysis will be performed on a sub-set of employees who respond affirmatively to a question, which inquires if participants have been diagnosed with one or more listed chronic conditions. The conditions increase the risk of complications from ARI/ILI or GI infections. The content in the measurement item to assess the number of ARI/ILI/GI infections has demonstrated acceptable validity and reliability in a previous study from a scale that does not have a formal title, utilized by Stedman-Smith, DuBois and Grey (2012). The scale measures whether or not participants have had self-reported (1) ARI/ILI or (2) GI infections using definitions from the CDC. Survey measurements will occur at baseline and weekly for 12 weeks. The number of self-reported infections during the 3-month trial will be counted, combined, and summed in the intervention and control groups; incidence rates and an incident rate ratio will be calculated with a 95% CI.
Improvement in Hygiene Behaviors as Self-Reported in Questionnaire | Approximately 90 days
  Survey items will be measured at the baseline; middle and conclusion of the study. Improvement in self-reported hand hygiene behaviors will be measured by a construct of seven items; the construct was part of a survey that does not have a formal title, which demonstrated acceptable validity and reliability from previous research by Stedman-Smith et al. (2012). The items contain a scale of 5 rankings from always (1) to never (5). Higher scores indicate more protective practices. Improvement in the use of hand sanitizer disinfectant wipes will be measured by a newly created item that measures the self-reported frequency of usage on a scale of 0-5, ranging from 2 or more times a day (5) to never (0). Higher scores indicate more protective self-reported hygiene practices. Mean scores will be calculated in the intervention group and in the control group and the two groups will be compared by mean differences.
Improvement in Hygiene-Related Attitudinal Beliefs as Self-Reported in Questionnaire | Approximately 90 days
  Measurement will occur at the baseline; middle and end of the study. Survey items measure constructs on a scale of 1-5 from strongly agree to strongly disagree: perceived beliefs about the benefits of performing protective hygiene behaviors; perceived employer and co-worker norms about hygiene behaviors; and perceived control beliefs about performing hygiene behaviors. Higher scores indicate stronger positive beliefs. Six of the nine constructs have demonstrated acceptable validity and reliability in a survey that does not have a formal title, created by Stedman-Smith et al. (2012). Three items were created regarding the use of disinfectant surface wipes and perceptions about environmental cleanliness. All survey items consist of a scale from 1-5, ranging from strongly agree (1) to strongly disagree (5). Higher scores indicate more positive beliefs. Mean scores will be calculated in the intervention and control groups, and mean differences will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Stedman-Smith, Ph.D., Principal Investigator — Kent State University, College of Public Health
Locations (1):
- The Golub Corporation (Price Chopper / Market 32), Schenectady, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The findings from the study will be published. The publication (s) will contain author contact information. Upon written request sent to the study PI, de-identified data that specifically pertains to the results that have been published will be shared through email.
  De-identified data that specifically pertains to the published results will be shared by email upon written request.
Supporting Information: SAP, Analytic Code
Time Frame: Study data will be available for one year following publication of the results.
Access Criteria: De-identified data that pertains to published results will be provided to other researchers by written request via email contact to the PI.

REFERENCES:
- [Background] Molinari NA, Ortega-Sanchez IR, Messonnier ML, Thompson WW, Wortley PM, Weintraub E, Bridges CB. The annual impact of seasonal influenza in the US: measuring disease burden and costs. Vaccine. 2007 Jun 28;25(27):5086-96. doi: 10.1016/j.vaccine.2007.03.046. Epub 2007 Apr 20. PMID 17544181
- [Background] Fendrick AM, Monto AS, Nightengale B, Sarnes M. The economic burden of non-influenza-related viral respiratory tract infection in the United States. Arch Intern Med. 2003 Feb 24;163(4):487-94. doi: 10.1001/archinte.163.4.487. PMID 12588210
- [Background] Baicker K, Cutler D, Song Z. Workplace wellness programs can generate savings. Health Aff (Millwood). 2010 Feb;29(2):304-11. doi: 10.1377/hlthaff.2009.0626. Epub 2010 Jan 14. PMID 20075081
- [Background] Boyce JM, Pittet D; Healthcare Infection Control Practices Advisory Committee. Society for Healthcare Epidemiology of America. Association for Professionals in Infection Control. Infectious Diseases Society of America. Hand Hygiene Task Force. Guideline for Hand Hygiene in Health-Care Settings: recommendations of the Healthcare Infection Control Practices Advisory Committee and the HICPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. Infect Control Hosp Epidemiol. 2002 Dec;23(12 Suppl):S3-40. doi: 10.1086/503164. PMID 12515399
- [Background] World Health Organization Writing Group; Bell D, Nicoll A, Fukuda K, Horby P, Monto A, Hayden F, Wylks C, Sanders L, van Tam J. Non-pharmaceutical interventions for pandemic influenza, national and community measures. Emerg Infect Dis. 2006 Jan;12(1):88-94. doi: 10.3201/eid1201.051371. PMID 16494723
- [Background] Centers for Disease Control and Prevention. Key facts about seasonal flu vaccine. Updated October 30, 2017: https://www.cdc.gov/flu/protect/keyfacts
- [Background] Aiello AE, Coulborn RM, Perez V, Larson EL. Effect of hand hygiene on infectious disease risk in the community setting: a meta-analysis. Am J Public Health. 2008 Aug;98(8):1372-81. doi: 10.2105/AJPH.2007.124610. Epub 2008 Jun 12. PMID 18556606
- [Background] Hubner NO, Hubner C, Wodny M, Kampf G, Kramer A. Effectiveness of alcohol-based hand disinfectants in a public administration: impact on health and work performance related to acute respiratory symptoms and diarrhoea. BMC Infect Dis. 2010 Aug 24;10:250. doi: 10.1186/1471-2334-10-250. PMID 20735818
- [Background] Savolainen-Kopra C, Haapakoski J, Peltola PA, Ziegler T, Korpela T, Anttila P, Amiryousefi A, Huovinen P, Huvinen M, Noronen H, Riikkala P, Roivainen M, Ruutu P, Teirila J, Vartiainen E, Hovi T. Hand washing with soap and water together with behavioural recommendations prevents infections in common work environment: an open cluster-randomized trial. Trials. 2012 Jan 16;13:10. doi: 10.1186/1745-6215-13-10. PMID 22243622
- [Background] Stedman-Smith M, DuBois CL, Grey SF, Kingsbury DM, Shakya S, Scofield J, Slenkovich K. Outcomes of a pilot hand hygiene randomized cluster trial to reduce communicable infections among US office-based employees. J Occup Environ Med. 2015 Apr;57(4):374-80. doi: 10.1097/JOM.0000000000000421. PMID 25719534
- [Background] Arbogast JW, Moore-Schiltz L, Jarvis WR, Harpster-Hagen A, Hughes J, Parker A. Impact of a Comprehensive Workplace Hand Hygiene Program on Employer Health Care Insurance Claims and Costs, Absenteeism, and Employee Perceptions and Practices. J Occup Environ Med. 2016 Jun;58(6):e231-40. doi: 10.1097/JOM.0000000000000738. PMID 27281645
- [Background] Centers for Disease Control and Prevention. How flu spreads. Updated October 5, 2017: https://www.cdc.gov/flu/about/index.html
- [Background] Stedman-Smith M, DuBois CL, Grey SF. Hand hygiene performance and beliefs among public university employees. J Health Psychol. 2015 Oct;20(10):1263-74. doi: 10.1177/1359105313510338. Epub 2013 Nov 20. PMID 24265297